CLINICAL TRIAL: NCT00336245
Title: A Randomized Trial of IUD Versus Hormonal Contraception in HIV-infected Women in Zambia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: Elizabeth Glaser Pediatric AIDS Foundation (Other); United States Agency for International Development (USAID) (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: EGPAF PG-51161
Record Dates: First submitted 2006-06-11; First posted 2006-06-13 (Estimated); Last update posted 2015-03-06 (Estimated); Status verified 2009-08

CONDITIONS: Pregnancy; HIV Infection
Keywords: Contraception; Women; HIV/AIDS; IUD; IUCD
MeSH Terms: conditions — HIV Infections; Acquired Immunodeficiency Syndrome | interventions — Hormonal Contraception

ARMS (2):
- Copper T Intrauterine Contraceptive Device (Experimental)
  Interventions: Device: Copper T Intrauterine Contraceptive Device
- Hormonal Contraception (Active Comparator)
  Interventions: Drug: Hormonal Contraception

INTERVENTIONS:
Device: Copper T Intrauterine Contraceptive Device
  Arms: Copper T Intrauterine Contraceptive Device
Drug: Hormonal Contraception
  Arms: Hormonal Contraception

SUMMARY:
A randomized trial of the intrauterine contraceptive device (IUD) versus user's choice hormonal contraception (injectable progestins or oral contraceptive pills) among HIV-infected, recently post-partum women in Lusaka, Zambia.

DETAILED DESCRIPTION:
In the year 2000, there were over 37, 000 new acceptors of family planning in the Lusaka District Clinics. A variety of methods were prescribed, including combined oral contraceptive pills, injectable progestins, the intrauterine copper device, condoms, and others. The most recent sentinel survey of reproductive age women estimated that approximately 30% of reproductive age women in Lusaka are HIV-infected. Since voluntary HIV counseling and testing is not yet universally available in many of the district clinics, women receive all different types of contraception regardless of their HIV status.

There is some observational data published recently that suggests hormonal contraception may increase HIV viral load in the female genital tract and potentially increase HIV transmission to the male partner. By contrast, barrier methods have historically been very unpopular in stable couples and are not used consistently in many cases despite intensive counseling. The IUCD represents one of the most inexpensive and effective methods of birth control available in Lusaka. However, it has not been studied adequately to make policy recommendations regarding its use in HIV infected women. The purpose of this study will be to evaluate safety and acceptability of the IUCD versus hormonal methods of contraception in HIV-infected and uninfected women in Lusaka. Specifically, we will 1) compare the contraceptive effectiveness of the IUCD to the standard practices of user-chosen hormonal contraception, 2) compare the rates of pelvic infection between IUD and hormonal contraceptive users, and 3) compare rates of method discontinuation.

Patients who have a continuing second trimester pregnancy, serologically confirmed HIV infection, a desire for 24 months of contraception, and a willingness to be randomly assigned either an IUCD or hormonal contraception postpartum will be screened at 32 weeks in their pregnancies to receive either an IUCD or user chosen hormonal contraception postpartum. Women will then be seen at postpartum weeks 4-6 for method randomization and then at months 6, 12, 18 and 24 to monitor pregnancy, continuation of method, side effects and any other problems. Women will be encouraged to return for problems at any time. At least once yearly, women will have a complete physical exam. CD4 and HIV clinical status will be monitored regularly.

ELIGIBILITY:
Inclusion Criteria:

* desire for at least 2 years of continuous contraception
* two or fewer sexual partners in the prior year

Exclusion Criteria:

* advanced HIV disease (WHO Stage III or IV)
* history of a bleeding disorder
* history of PID within the prior five years
* less than 16 years of age (the "age of majority" in Zambia).

Min Age: 16 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 600
Dates: Start 2002-06; Primary Completion 2005-10 (Actual); Study Completion 2005-10 (Actual)

PRIMARY OUTCOMES:
Incident pregnancy

SECONDARY OUTCOMES:
Safety
Method discontinuation rates

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Stringer, MD, Principal Investigator — University of Alabama at Birmingham